CLINICAL TRIAL: NCT00924456
Title: A Randomized Controlled Trial of the Transcendental Meditation Program on Blood Pressure, Psychological Distress, and Coping in Young Adults
Brief Title: A Clinical Trial of the Transcendental Meditation (TM) Program on Blood Pressure, Psychological Distress, and Coping
Acronym: AU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maharishi International University (Other)
Collaborators: American University (Other); Abramson Family Foundation (Other)
Responsible Party: Principal Investigator, Robert Schneider, MD, Director and Dean, Maharishi International University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: AF-0001
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: High-normal Blood Pressure; Psychological Stress
Keywords: Transcendental Meditation; blood pressure; psychological distress; high psychological distress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcendental Meditation program (Experimental): a natural effortless mental technique practiced sitting quietly 20 minutes twice a day
  Interventions: Behavioral: Transcendental Meditation program
- Wait list control (Placebo Comparator): student subjects on wait list control
  Interventions: Behavioral: Transcendental Meditation program

INTERVENTIONS:
Behavioral: Transcendental Meditation program — a natural effortless mental technique
  Other Names: TM

SUMMARY:
The purpose of this trial is to show that the Transcendental Meditation program can decrease blood pressure in young adults (college students) and is associated with decreased psychological distress and coping ability.

DETAILED DESCRIPTION:
Psychological distress contributes to the development of hypertension in young adults. This was a randomized controlled trial of 296 university students randomly allocated to either the Transcendental Meditation® program or wait-list control. At baseline and after three months posttest, systolic and diastolic blood pressure, psychological distress (total mood disturbance, anxiety, depression, anger/hostility) and coping ability (global constructive thinking) were measured.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* currently enrolled in an undergraduate or graduate program through August 2006

Exclusion Criteria:

* history of:

  * hypertension
  * hypoglycemia
  * chronic fainting
  * coronary heart disease
  * current systolic/diastolic blood pressure above 140/90 mm Hg or below 90/60 mm Hg

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2006-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
clinic systolic and diastolic blood pressure | 3 months

SECONDARY OUTCOMES:
psychological distress (anxiety, depression, anger/hostility) and coping (constructive thinking) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Schneider, M.D., Principal Investigator — Maharishi International University
Locations (1):
- American University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Nidich SI, Rainforth MV, Haaga DA, Hagelin J, Salerno JW, Travis F, Tanner M, Gaylord-King C, Grosswald S, Schneider RH. A randomized controlled trial on effects of the Transcendental Meditation program on blood pressure, psychological distress, and coping in young adults. Am J Hypertens. 2009 Dec;22(12):1326-31. doi: 10.1038/ajh.2009.184. Epub 2009 Oct 1. PMID 19798037
- [Result] Travis F, Haaga DA, Hagelin J, Tanner M, Nidich S, Gaylord-King C, Grosswald S, Rainforth M, Schneider RH. Effects of Transcendental Meditation practice on brain functioning and stress reactivity in college students. Int J Psychophysiol. 2009 Feb;71(2):170-6. doi: 10.1016/j.ijpsycho.2008.09.007. Epub 2008 Sep 30. PMID 18854202
- [Result] Haaga DA, Grosswald S, Gaylord-King C, Rainforth M, Tanner M, Travis F, Nidich S, Schneider RH. Effects of the Transcendental Meditation Program on Substance Use among University Students. Cardiol Res Pract. 2011 Mar 21;2011:537101. doi: 10.4061/2011/537101. PMID 21559213